CLINICAL TRIAL: NCT02687373
Title: Safety, Tolerability and Efficacy of PfSPZ Vaccine Administered by Direct Venous Inoculation (DVI) to Healthy Children and Infants 5 Months Through 9 Years of Age Living in an Area of High Malaria Transmission in Western Kenya: Age De-escalation and Dose Escalation and a Double Blind, Randomized Placebo-Controlled Trial for Safety and Efficacy
Brief Title: Safety, Tolerability and Efficacy of PfSPZ Vaccine in Healthy Children and Infants 5 Months - 9 Years Living in Kenya
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Kenya Medical Research Institute (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KEMRI/SERU/CGHR/017/3129; CDC IRB Protocol #6787 (Other: CDC, USA)
Record Dates: First submitted 2016-02-09; First posted 2016-02-22 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; PfSPZ Vaccine
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (30):
- Part 1: Grp 1A - PfSPZ Vaccine (Experimental): Children aged 5-9 years (inclusive) of age will be enrolled in this group.
  N=8; Dose of 4.5 x 10^5 PfSPZ Vaccine administered DVI, as a single vaccination.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 1A - Normal Saline (Placebo Comparator): Children aged 5-9 years (inclusive) of age will be enrolled in this group.
  N=4; Normal saline administered DVI, as a single vaccination.
  Interventions: Other: Normal Saline
- Part 1: Grp 1B - PfSPZ Vaccine (Experimental): Children aged 5-9 years (inclusive) of age will be enrolled in this group.
  N=8; Two doses of 9.0 x 10^5 PfSPZ Vaccine administered DVI, 8 weeks apart. The 1st dose will be administered 2 weeks after Grp 1A dose has been shown to be well-tolerated and without safety concerns. The 2nd dose will be administered 8 weeks after the 1st dose in this group does not show any safety signals.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 1B - Normal Saline (Placebo Comparator): Children aged 5-9 years (inclusive) of age will be enrolled in this group.
  N=4; Two doses of normal saline administered DVI, 8 weeks apart. The 1st dose will be administered 2 weeks after Grp 1A dose has been shown to be well-tolerated and without safety concerns. The 2nd dose will be administered 8 weeks after the 1st dose in this group does not show any safety signals.
  Interventions: Other: Normal Saline
- Part 1: Grp 1C - PfSPZ Vaccine (Experimental): Children aged 5-9 years (inclusive) of age will be enrolled in this group.
  N=8; Two doses of 1.8 x 10^6 PfSPZ Vaccine administered DVI, 8 weeks apart. The 1st dose will be administered 2 weeks after the 1st dose of Grp 1B has been shown to be well-tolerated and without safety concerns. The 2nd dose will be administered 8 weeks after the 1st dose in this group does not show any safety signals.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 1C - Normal Saline (Placebo Comparator): Children aged 5-9 years (inclusive) of age will be enrolled in this group.
  N=4; Two doses of normal saline administered DVI, 8 weeks apart. The 1st dose will be administered after the 1st dose of Grp 1B has been shown to be well-tolerated and without safety concerns. The 2nd dose will be administered 8 weeks after the 1st dose in this group does not show any safety signals.
  Interventions: Other: Normal Saline
- Part 1: Grp 2A - PfSPZ Vaccine (Experimental): Children aged 13-59 months (inclusive) of age will be enrolled in this group.
  N=8; Dose of 1.35 x 10^5 PfSPZ Vaccine administered DVI, as a single vaccination. This dose will be administered 2 weeks after the 1st dose of Grp 1B has been shown to be well-tolerated and without safety concerns.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 2A - Normal Saline (Placebo Comparator): Children aged 13-59 months (inclusive) of age will be enrolled in this group.
  N=4; Normal saline administered DVI, as a single vaccination. This dose will be administered 2 weeks after the 1st dose of Grp 1B has been shown to be well-tolerated and without safety concerns.
  Interventions: Other: Normal Saline
- Part 1: Grp 2B - PfSPZ Vaccine (Experimental): Children aged 13-59 months (inclusive) of age will be enrolled in this group.
  N=8; Dose of 2.7 x 10^5 PfSPZ Vaccine administered DVI, as a single vaccination. This dose will be administered 2 weeks after Grp 2A has been shown to be well-tolerated and without safety concerns.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 2B - Normal Saline (Placebo Comparator): Children aged 13-59 months (inclusive) of age will be enrolled in this group.
  N=4; Normal saline administered DVI, as a single vaccination. This dose will be administered 2 weeks after Grp 2A has been shown to be well-tolerated and without safety concerns.
  Interventions: Other: Normal Saline
- Part 1: Grp 2C - PfSPZ Vaccine (Experimental): Children aged 13-59 months (inclusive) of age will be enrolled in this group.
  N=8; Dose of 4.5 x 10^5 PfSPZ Vaccine administered DVI, as a single vaccination. This dose will be administered 2 weeks after Grp 2B has been shown to be well-tolerated and without safety concerns.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 2C - Normal Saline (Placebo Comparator): Children aged 13-59 months (inclusive) of age will be enrolled in this group.
  N=4; Normal saline administered DVI, as a single vaccination. This dose will be administered 2 weeks after Grp 2B has been shown to be well-tolerated and without safety concerns.
  Interventions: Other: Normal Saline
- Part 1: Grp 2D - PfSPZ Vaccine (Experimental): Children aged 13-59 months (inclusive) of age will be enrolled in this group.
  N=8; Two doses of 9.0 x 10^5 PfSPZ Vaccine administered DVI, 8 weeks apart. The 1st dose will be administered 2 weeks after Grp 2C has been shown to be well-tolerated and without safety concerns. The 2nd dose will be administered 8 weeks after the 1st dose in this group does not show any safety signals.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 2D - Normal Saline (Placebo Comparator): Children aged 13-59 months (inclusive) of age will be enrolled in this group.
  N=4; Two doses of normal saline administered DVI, 8 weeks apart. The 1st dose will be administered 2 weeks after Grp 2C has been shown to be well-tolerated and without safety concerns. The 2nd dose will be administered 8 weeks after the 1st dose in this group does not show any safety signals.
  Interventions: Other: Normal Saline
- Part 1: Grp 2E - PfSPZ Vaccine (Experimental): Children aged 13-59 months (inclusive) of age will be enrolled in this group.
  N=8; Two doses of 1.8 x 10^6 PfSPZ Vaccine administered DVI, 8 weeks apart. The 1st dose will be administered 2 weeks after Grp 2D has been shown to be well-tolerated and without safety concerns. The 2nd dose will be administered 8 weeks after the 1st dose in this group does not show any safety signals.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 2E - Normal Saline (Placebo Comparator): Children aged 13-59 months (inclusive) of age will be enrolled in this group.
  N=4; Two doses of normal saline administered DVI, 8 weeks apart. The 1st dose will be administered 2 weeks after Grp 2D has been shown to be well-tolerated and without safety concerns. The 2nd dose will be administered 8 weeks after the 1st dose in this group does not show any safety signals.
  Interventions: Other: Normal Saline
- Part 1: Grp 3A - PfSPZ Vaccine (Experimental): Children aged 5-12 months (inclusive) of age will be enrolled in this group.
  N=8; Dose of 1.35 x 10^5 PfSPZ Vaccine administered DVI, as a single vaccination. This dose will be administered 2 weeks after Grp 2B has been shown to be well-tolerated and without safety concerns.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 3A - Normal Saline (Placebo Comparator): Children aged 5-12 months (inclusive) of age will be enrolled in this group.
  N=4; Normal saline administered DVI, as a single vaccination. This dose will be administered 2 weeks after Grp 2B has been shown to be well-tolerated and without safety concerns.
  Interventions: Other: Normal Saline
- Part 1: Grp 3B - PfSPZ Vaccine (Experimental): Children aged 5-12 months (inclusive) of age will be enrolled in this group.
  N=8; Dose of 2.7 x 10^5 PfSPZ Vaccine administered DVI, as a single vaccination. This dose will be administered 2 weeks after Grp 3A has been shown to be well-tolerated and without safety concerns.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 3B - Normal Saline (Placebo Comparator): Children aged 5-12 months (inclusive) of age will be enrolled in this group.
  N=4; Normal saline administered DVI, as a single vaccination. This dose will be administered 2 weeks after Grp 3A has been shown to be well-tolerated and without safety concerns.
  Interventions: Other: Normal Saline
- Part 1: Grp 3C - PfSPZ Vaccine (Experimental): Children aged 5-12 months (inclusive) of age will be enrolled in this group.
  N=8; Dose of 4.5 x 10^5 PfSPZ Vaccine administered DVI, as a single vaccination. This dose will be administered 2 weeks after Grp 3B has been shown to be well-tolerated and without safety concerns.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 3C - Normal Saline (Placebo Comparator): Children aged 5-12 months (inclusive) of age will be enrolled in this group.
  N=4; Normal saline administered DVI, as a single vaccination. This dose will be administered 2 weeks after Grp 3B has been shown to be well-tolerated and without safety concerns.
  Interventions: Other: Normal Saline
- Part 1: Grp 3D - PfSPZ Vaccine (Experimental): Children aged 5-12 months (inclusive) of age will be enrolled in this group.
  N=8; Two doses of 9.0 x 10^5 PfSPZ Vaccine administered DVI, 8 weeks apart. The 1st dose will be administered 2 weeks after Grp 3C has been shown to be well-tolerated and without safety concerns. The 2nd dose will be administered 8 weeks after the 1st dose in this group does not show any safety signals.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 3D - Normal Saline (Placebo Comparator): Children aged 5-12 months (inclusive) of age will be enrolled in this group.
  N=4; Two doses of normal saline administered DVI, 8 weeks apart. The 1st dose will be administered 2 weeks after Grp 3C has been shown to be well-tolerated and without safety concerns. The 2nd dose will be administered 8 weeks after the 1st dose in this group does not show any safety signals.
  Interventions: Other: Normal Saline
- Part 1: Grp 3E - PfSPZ Vaccine (Experimental): Children aged 5-12 months (inclusive) of age will be enrolled in this group.
  N=8; Two doses of 1.8 x 10^6 PfSPZ Vaccine administered DVI, 8 weeks apart. The 1st dose will be administered 2 weeks after Grp 3D has been shown to be well-tolerated and without safety concerns. The 2nd dose will be administered 8 weeks after the 1st dose in this group does not show any safety signals.
  Interventions: Biological: PfSPZ Vaccine
- Part 1: Grp 3E - Normal Saline (Placebo Comparator): Children aged 5-12 months (inclusive) of age will be enrolled in this group.
  N=4; Two doses of normal saline administered DVI, 8 weeks apart. The 1st dose will be administered 2 weeks after Grp 3D has been shown to be well-tolerated and without safety concerns. The 2nd dose will be administered 8 weeks after the 1st dose in this group does not show any safety signals.
  Interventions: Other: Normal Saline
- Part 2: Group 1 - PfSPZ Vaccine (Experimental): Infants aged 5-12 months (inclusive) of age at vaccination will be enrolled in Part 2.
  N=104; the highest dose that is determined to be safe and well tolerated in the Part 1 trial, administered in 3 doses by DVI at 0, 8 and 16 weeks. Likely dosage will be 1.8 x 10^6 PfSPZ per dose.
  Interventions: Biological: PfSPZ Vaccine
- Part 2: Group 2 - PfSPZ Vaccine (Experimental): Infants aged 5-12 months (inclusive) of age at vaccination will be enrolled in Part 2.
  N=104; the second highest dose, which is half of the highest dose, administered in 3 doses by DVI at 0, 8 and 16 weeks. Likely dosage will be 9.0 x 10^5 PfSPZ per dose.
  Interventions: Biological: PfSPZ Vaccine
- Part 2: Group 3 - PfSPZ Vaccine (Experimental): Infants aged 5-12 months (inclusive) of age at vaccination will be enrolled in Part 2.
  N=104; a lower dose (half of the second highest dose) administered in 3 doses by DVI at 0, 8, 16 weeks. Likely dosage will be 4.5x 10^5 PfSPZ per dose.
  Interventions: Biological: PfSPZ Vaccine
- Part 2: Group 4 - Normal Saline (Placebo Comparator): Infants aged 5-12 months (inclusive) of age at vaccination will be enrolled in Part 2.
  N=104; a placebo arm, will receive normal saline by DVI, 3 times at 8 week intervals.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: PfSPZ Vaccine — Aseptic, purified, cryopreserved, radiation-attenuated Plasmodium falciparum sporozoites
  Arms: Part 1: Grp 1A - PfSPZ Vaccine; Part 1: Grp 1B - PfSPZ Vaccine; Part 1: Grp 1C - PfSPZ Vaccine; Part 1: Grp 2A - PfSPZ Vaccine; Part 1: Grp 2B - PfSPZ Vaccine; Part 1: Grp 2C - PfSPZ Vaccine; Part 1: Grp 2D - PfSPZ Vaccine; Part 1: Grp 2E - PfSPZ Vaccine; Part 1: Grp 3A - PfSPZ Vaccine; Part 1: Grp 3B - PfSPZ Vaccine; Part 1: Grp 3C - PfSPZ Vaccine; Part 1: Grp 3D - PfSPZ Vaccine; Part 1: Grp 3E - PfSPZ Vaccine; Part 2: Group 1 - PfSPZ Vaccine; Part 2: Group 2 - PfSPZ Vaccine; Part 2: Group 3 - PfSPZ Vaccine
Other: Normal Saline — 0.9% Sodium chloride
  Arms: Part 1: Grp 1A - Normal Saline; Part 1: Grp 1B - Normal Saline; Part 1: Grp 1C - Normal Saline; Part 1: Grp 2A - Normal Saline; Part 1: Grp 2B - Normal Saline; Part 1: Grp 2C - Normal Saline; Part 1: Grp 2D - Normal Saline; Part 1: Grp 2E - Normal Saline; Part 1: Grp 3A - Normal Saline; Part 1: Grp 3B - Normal Saline; Part 1: Grp 3C - Normal Saline; Part 1: Grp 3D - Normal Saline; Part 1: Grp 3E - Normal Saline; Part 2: Group 4 - Normal Saline

SUMMARY:
This study will be conducted in Siaya County in Nyanza Province, western Kenya. Healthy children aged 5 months through 9 years of age living within approximately 10 km of the study clinic(s) (Siaya County Referral Hospital, or Wagai dispensary, a government health facility in Wagai division) will be eligible for participation in Part 1; healthy infants aged 5 months - 12 months inclusive will be eligible for Part 2.

DETAILED DESCRIPTION:
Part 1: Age De-Escalation and Dose Escalation Part 1 of this trial is a randomized blinded evaluation of the safety and tolerability of PfSPZ Vaccine administered by DVI in healthy children and infants living in an area of high malaria transmission. A maximum of 156 children from 5 months to 9 years inclusive at vaccination will be enrolled and randomized to receive vaccine or normal saline (NS) placebo by DVI. Total participation time in the dose escalation trial ranges from 5-16 weeks per participant from screening visit to close out or 4 - 12 weeks from enrolment to close out.

Vaccination will begin in the 5-9 year age group at a dosage of 4.5 x10^5 PfSPZ. A single vaccination will be administered by DVI to each of 12 participants aged 5-9 years (inclusive) of age, 8 receiving PfSPZ vaccine and 4 participants receiving NS placebo by DVI, with treatment allocation randomized and double-blind. Once the initial dose has been shown to be well tolerated and without safety concerns, the next higher dose of 9.0 x 10^5 PfSPZ will be administered to a second group of 5-9 year olds. Once this has been shown to be well tolerated and without safety concerns, the highest dose of 1.8 x 10^6 PfSPZ will be given to a third group of 5-9 year olds and concurrently the lowest dose (1.35 x10^5) will be given to a same-sized group of younger children aged 13-59 months. Two weeks later, this dose will be escalated to 2.7 x10^5 PfSPZ in a second group of children aged 13-59 months. Only once this dose is shown to be well-tolerated and without safety concerns will PfSPZ Vaccine, at the lowest dose, be given to infants aged 5 - 12 months. Within each age group, dosages will increase stepwise until they reach 1.8 x 10^6 PfSPZ, with the initiation of each group staggered by at least 2 weeks, provided that no safety thresholds are surpassed. In each dosage level, the PfSPZ Vaccine or placebo will be provided to a limited number of participants each day (e.g. 3 participants from one age group on days 1 through 4). The PfSPZ Vaccine dose will only be increased to the next dose level when safety has been assessed in subjects of the first group. The same procedures will be followed for all doses. Children in all age groups who are enrolled to receive the 2 highest doses, i.e. 9.0 x 10^5 or 1.8 x 10^6 PfSPZ, or placebo, will receive a second vaccination of the same dose after 8 weeks, provided the first vaccination at this dose level did not show safety signals.

Part 2: Safety and Efficacy Part of this study will be conducted in the outpatient areas of Siaya County Referral Hospital, a large referral hospital in western Kenya and in Wagai dispensary. A maximum of 416 infants from 5 M to 12 M inclusive at vaccination will be enrolled into this safety and efficacy trial and randomized to receive PfSPZ Vaccine at a dose determined during Part 1 of the trial (dose escalation), but likely to be 4.5x10^5, 9.0 x10^5and 1.8 x 10^6 administered x 3 doses ; and NS placebo administered x 3 doses, all by DVI administered at 8 week intervals.

Participants (N = 416, with 104 in each study arm) will be randomly assigned in a double blinded fashion to receive one of the following PfSPZ Vaccine regimes:

Group 1 (N=104): The highest dose that is determined to be safe and well tolerated in the Part 1 trial, administered in 3 doses by DVI at 0, 8 and 16 weeks. Likely dosage will be 1.8 x 10^6 PfSPZ per dose.

Group 2 (N=104): The second highest dose, which is half of the highest dose, administered in 3 doses by DVI at 0, 8 and 16 weeks. Likely dosage will be 9.0 x 10^5 PfSPZ per dose.

Group 3 (N=104): A lower dose (half of the second highest dose) administered in 3 doses by DVI at 0, 8, 16 weeks. Likely dosage will be 4.5x 10^5 PfSPZ per dose.

Group 4 (N=104): A placebo arm, will receive NS by DVI, 3 times at 8 week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children 5 months - 9 years inclusive (Part 1) and healthy infants 5-12 months inclusive (Part 2)
* HIV negative
* Able to participate for the duration of the study.
* Parents/guardians over the age of 18 years able and willing to provide informed consent/permission. The consent/permission will be in writing. For adult parents or guardians who are illiterate, an impartial witness can sign the consent/permission form on behalf of the parent and the parent/guardian will provide a thumb print.

Exclusion Criteria:

* Positive HIV test or breastfeeding infants or children of a known HIV positive mother (per Kenyan guidelines, these HIV exposed breastfeeding children should be on cotrimoxazole)
* Refusal of HIV testing
* Elevated ALT (liver function test) ≥2x ULN ( ALT >84 U/L)
* Abnormal hematological parameters defined as: hemoglobin < 8 g/dl, WBC <1500 / mm3, neutrophils <750/ mm3, platelet count <75.000/ mm3
* Abnormal renal function test with creatinine >0.9 mg/dL
* Known sickle cell disease and other inherited blood cell disorders like thalassemia and G6PD deficiency
* Current use of systemic immunosuppressant pharmacotherapy
* Current significant medical condition (cardiac, hepatic, renal, or hematological) or evidence of any other serious underlying medical condition identified by medical history, physical examination, or laboratory examination
* History of a splenectomy
* History of neurologic disorder (including seizures, other than uncomplicated febrile seizures)
* Known allergy to any component of the vaccine formulation, history of anaphylactic response to mosquito-bites, or known allergy to first or second line anti-malarials used to treat malaria
* Plan to participate in another investigational vaccine/drug research during or within 1 month of this study end
* Prior participation in a malaria vaccine trial
* Participation in the PfSPZ Vaccine Trial Part 1 (for Part 2 only)
* History of any other illness or condition which, in the investigator's judgment, may substantially increase the risk associated with the subject's participation in the protocol or compromise the scientific objectives
* Child/orphan in institutional care

Ages: 5 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 337 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Part 1 - Incidence and type of adverse events (AE) | Collected from day of each vaccination until day 28 post vaccination
  Incidence and type of solicited and unsolicited adverse events including breakthrough malaria infections and clinical laboratory assessments (hematological, liver and renal function) will be collected within 28 days after each vaccination. Proportions of participants with AEs and frequencies of individual AEs will be calculated and compared against participants in the same age category and dose group receiving placebo.
Part 1 - Incidence and type of possibly/probably or definitely related serious adverse events (SAEs) | Collected from day of first vaccination until close out visit (28 days for 3 lower doses, 84 days for 2 higher doses)
  Incidence of all hospitalizations, deaths, disabilities caused by at least possibly related SAEs during study participation
Part 1 - Assessment of Pf-specific antibodies in the different age categories and to the different vaccine doses | Collected 1 week after each vaccination
  Collection of blood samples for antibodies on day 8 after each vaccination. Following vaccination serum will be taken and an assessment of Plasmodium falciparum (Pf)f-specific antibodies against specific malaria proteins such as the circumsporozoite protein (CSP) PfCSP and whole Pf sporozoites (SPZ) will be determined by enzyme-linked immunosorbent assay (ELISA) and automated immunofluorescence assay (aIFA) respectively.
Part 2 - Incidence and type of adverse events in infants 5-12 months of age following administration of PfSPZ Vaccine | Collected from day of each vaccination until day 28 post vaccination
  Incidence and type of solicited and unsolicited adverse events including breakthrough malaria infections and clinical laboratory assessments (hematological, liver and renal function) will be collected during 28 days after each vaccination.
Part 2 - Incidence and type of possibly/probably or definitely related serious adverse events (SAEs) following administration of PfSPZ Vaccine | Collected from day of first vaccination through the 12-month follow-up period.
  Incidence of all hospitalizations, deaths, disabilities caused by at least possibly related to the study product during the 12-month follow-up period.
Part 2 - Assessment of Pf-specific antibodies in infants of 5-12 months to three vaccinations of PfSPZ Vaccine | Collected 1 week after the first and second vaccination and 2 weeks after the third vaccination.
  Collection of blood samples for antibodies on day 8 after vaccination 1 and 2 and day 15 after the third PfSPZ vaccination. Following vaccination serum will be taken and an assessment of Plasmodium falciparum (Pf)f-specific antibodies against specific malaria proteins such as the circumsporozoite protein (CSP) PfCSP and whole Pf sporozoites (SPZ) will be determined by enzyme-linked immunosorbent assay (ELISA) and automated immunofluorescence assay (aIFA) respectively.
Part 2 - Ratio of Pf positive blood smear (+BS) in experimental arm to Pf +BS in placebo arm to determine efficacy of PfSPZ Vaccine during 6 months after last dose | 2 weeks to 6 months after the last vaccine dose
  Efficacy against malaria infection of PfSPZ Vaccine administered to infants 5-12 months of age in 3 doses by passive and active surveillance for naturally acquired Pf infection, measured by blood smear microscopy, during 6 months following the last vaccine dose.

SECONDARY OUTCOMES:
Part 2 - Ratio of Pf +BS in experimental arm to Pf +BS in placebo arm to determine efficacy of PfSPZ Vaccine during 12 months after last dose | 2 weeks to 12 months after the last vaccine dose
  Efficacy against malaria of PfSPZ Vaccine administered to infants 5-12 months of age in 3 doses by passive and active surveillance for naturally acquired Pf infection, measured by blood smear microscopy, during 12 months following the last vaccine dose will be performed and the prevalence ratio of the prevalence of malaria infection by blood smear between each dose study arm and placebo will be compared.
Part 2 - Ratio of Pf positive PCR in experimental arm to Pf positive PCR in placebo arm to determine efficacy against submicroscopic malaria infection of PfSPZ Vaccine following 6 and 12 months after the last dose | 2 weeks to 6 and 12 months after the last vaccine dose
  Efficacy against submicroscopic malaria infection of PfSPZ Vaccine administered to infants 5-12 months of age in 3 doses by passive and active surveillance for naturally acquired Pf infection, measured by PCR, during 6 and 12 months following the last vaccine dose.
Part 2 - Assessment of Pf-specific antibodies, parasite-specific T cell responses and RNA sequencing. | Before the first vaccination, 1 week after vaccination 1 and 2, 2 weeks after vaccination 3 and at 6 months and 12 months after the last vaccination
  Collection of blood samples for Anti PfSPZ antibodies and RNA sequencing at different time points. Following vaccination serum will be taken and an assessment of Plasmodium falciparum (Pf)f-specific antibodies against specific malaria proteins such as the circumsporozoite protein (CSP) PfCSP and whole Pf sporozoites (SPZ) will be determined by enzyme-linked immunosorbent assay (ELISA) and automated immunofluorescence assay (aIFA). For assessment of parasite-specific T cell responses, PBMCs will be assessed by multi-parameter flow cytometry and / or ELISPOT, and intracellular cytokine staining. RNA sequencing from whole blood will be performed by processing the RNA and performing deep sequencing. Analysis of gene expression will be performed to develop biomarkers and predictors of protection.
Part 2 - Assessment of Pf-specific antibodies, parasite-specific T cell responses and RNA sequencing to determine correlation of immune response with efficacy | Entire study period
  Comparison of the immune response at different time points and the protection against naturally acquired Pf infection. Following vaccination serum will be taken and an assessment of Plasmodium falciparum (Pf)f-specific antibodies against specific malaria proteins such as the circumsporozoite protein (CSP) PfCSP and whole Pf sporozoites (SPZ) will be determined by enzyme-linked immunosorbent assay (ELISA) and automated immunofluorescence assay (aIFA). For assessment of parasite-specific T cell responses, PBMCs will be assessed by multi-parameter flow cytometry and / or ELISPOT, and intracellular cytokine staining. RNA sequencing from whole blood will be performed by processing the RNA and performing deep sequencing. Analysis of gene expression will be performed to develop biomarkers and predictors of protection.

OTHER OUTCOMES:
Ratio of Pf +BS in experimental arm to Pf +BS in placebo arm to determine efficacy against Pf infection at certain parasite thresholds in each study arm | 2 weeks to 12 months after last vaccination
  Passive and active surveillance for naturally acquired Pf infection, measured by blood smear microscopy, during 12 months following the last dose in each study arm will be performed and the Pf infection by blood smear at parasite density >400 or >5000 parasites per microliter between each dose study arm and placebo will be compared.
Ratio of Pf +BS in experimental arm to Pf +BS in placebo arm to determine efficacy against clinical malaria and malaria hospitalization in each study arm | 2 weeks to 12 months after last vaccination
  Passive and active surveillance for naturally acquired Pf infection of > 5000 parasites per microliter measured by blood smear microscopy associated with fever (clinical malaria) and/or hospitalization as well as hospitalization for severe malarial anemia, during 12 months following the last dose in each study arm will be performed and each study arm will be compared with the placebo group.
Effect of vaccination on anemia | 6 months and 12 months after last vaccination
  Measure hemoglobin at 6 months and 12 months after the last vaccination and compare hemoglobin levels in each study arm with the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Oneko, MD, Principal Investigator — Kenya Medical Research Institute, Centre for Global Health Research, Kisumu, Kenya
Locations (1):
- Center for Global Health Research, KEMRI, Kisian, Siaya County, Kenya

REFERENCES:
- [Derived] Oneko M, Steinhardt LC, Yego R, Wiegand RE, Swanson PA, Kc N, Akach D, Sang T, Gutman JR, Nzuu EL, Dungani A, Kim Lee Sim B, Oloo PN, Otieno K, Bii DK, Billingsley PF, James ER, Kariuki S, Samuels AM, Jongo S, Chebore W, Abdulla S, Daubenberger C, Mpina M, Styers D, Potter GE, Abarbanell G, Richie TL, Hoffman SL, Seder RA. Safety, immunogenicity and efficacy of PfSPZ Vaccine against malaria in infants in western Kenya: a double-blind, randomized, placebo-controlled phase 2 trial. Nat Med. 2021 Sep;27(9):1636-1645. doi: 10.1038/s41591-021-01470-y. Epub 2021 Sep 13. PMID 34518679
- [Derived] Oneko M, Cherop YR, Sang T, Gutman JR, Wiegand R, Nyang'au EM, Odila AD, Akach D, Hamel MJ, Samuels AM, Kariuki S, Abebe Y, Nzuu EL, Wijayalath W, James ER, Sim BKL, Billingsley PF, Richie TL, Hoffman SL, Seder RA, Steinhardt LC. Feasibility of direct venous inoculation of the radiation-attenuated Plasmodium falciparum whole sporozoite vaccine in children and infants in Siaya, western Kenya. Vaccine. 2020 Jun 15;38(29):4592-4600. doi: 10.1016/j.vaccine.2020.05.008. Epub 2020 May 19. PMID 32444192
- [Derived] Steinhardt LC, Richie TL, Yego R, Akach D, Hamel MJ, Gutman JR, Wiegand RE, Nzuu EL, Dungani A, Kc N, Murshedkar T, Church LWP, Sim BKL, Billingsley PF, James ER, Abebe Y, Kariuki S, Samuels AM, Otieno K, Sang T, Kachur SP, Styers D, Schlessman K, Abarbanell G, Hoffman SL, Seder RA, Oneko M. Safety, Tolerability, and Immunogenicity of Plasmodium falciparum Sporozoite Vaccine Administered by Direct Venous Inoculation to Infants and Young Children: Findings From an Age De-escalation, Dose-Escalation, Double-blind, Randomized Controlled Study in Western Kenya. Clin Infect Dis. 2020 Aug 14;71(4):1063-1071. doi: 10.1093/cid/ciz925. PMID 31555824